CLINICAL TRIAL: NCT07074522
Title: Transvaginal Ultrasound Assessment of Caesarean Section Uterine Scar Closed by Single Versus Double Layer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Said Abd El Kareem Said Saad, Resident of Obstetrics and Gynecology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS426/11/23
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Transvaginal Ultrasound; Caesarean Section; Uterine Scar; Single Layer; Double Layer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single layer group (Experimental): Patients who underwent single-layer closure of the transverse lower segment during cesarean section.
  Interventions: Procedure: Single-layer closure
- Double layer group (Experimental): Patients who underwent double-layer closure of the transverse lower segment during cesarean section.
  Interventions: Procedure: Double-layer closure

INTERVENTIONS:
Procedure: Single-layer closure — Patients who underwent single-layer closure of the transverse lower segment during cesarean section.
  Arms: Single layer group
Procedure: Double-layer closure — Patients who underwent double-layer closure of the transverse lower segment during cesarean section.
  Arms: Double layer group

SUMMARY:
This study aimed to evaluate uterine scar thickness and integrity using transvaginal ultrasonography in women randomly assigned to single versus double-layer closure of the uterine incision, with a comparison between the two groups.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most commonly performed major abdominal operations in women in both high and low-income countries.

Single-layer closure using a running locking stitch is associated with decreased operative time and fewer additional haemostasis sutures. An extensive Canadian study found a fourfold increase in the risk of uterine rupture in a woman who had a single layer in their previous pregnancy.

Transvaginal ultrasound is a validated tool for evaluating uterine scar defects, commonly referred to as a niche. It is used to asses the uterine scar thickness in a women with previous cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 40 years old.
* Pregnant women underwent their first cesarean section.

Exclusion Criteria:

* Body mass index (BMI) ≥ 30 kg /m2.
* Multiple gestations.
* Uterine malformation.
* Placenta previa.
* Placenta accreta.
* Uterine or cervical fibroid.
* Any previous uterine operation or any medical disease that compromises wound healing, such as diabetes mellitus, collagen diseases, anemia, or corticosteroid therapy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women underwent their first cesarean section.
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Uterine scar thickness | 6 months postoperatively
  Uterine scar thickness was evaluated by transvaginal ultrasound six weeks, three months, and six months postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.